CLINICAL TRIAL: NCT00698113
Title: Parent-Delivered Massage in Paediatric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centennial College (Other)
Collaborators: SickKids Foundation (Other); Stollery Children's Hospital (Other); Canadian Institute of Natural and Integrative Medicine (Other)
Responsible Party: Trish Dryden, RMT, M.Ed, Director, Applied Research Centre, Centennial College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CENT-SK-CAM07-323R; CAM 07-323R
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Anxiety; Depression; Stress; Pediatric Cancers
Keywords: anxiety; depression; stress; cancer symptoms; pediatric cancer; massage; parent delivered massage
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms | interventions — Massage; Microscopy, Interference

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): This group receives the massage intervention for a period of six weeks. Children and parents are asked to journal weekly for the six week period.
  Interventions: Procedure: Massage; Other: Journaling
- 2 (No Intervention): The control group does not receive any massage intervention during the initial six weeks of the study. The children are asked to journal during this six week period.
  Interventions: Other: Journaling

INTERVENTIONS:
Procedure: Massage — Children will receive a 10-15 minute massage seated (clothed), or in bed (clothed or unclothed) each day using the following protocol: stroking, effleurage, petrissage, muscle squeezing, effleurage, stroking. Massaged areas can include the back, arms and legs.
  Parents will receive a one hour educational session with a Massage Therapist, a DVD, and written materials that all illustrate the required protocol.
  Other Names: massage therapy
  Arms: 1
Other: Journaling — Children will complete weekly journals about their feelings. These journals will either be drawn or written based on the preference of the child. Parents will complete a weekly journal outlining the number of massages given to their child, barriers that prevented massage, and their experience of giving the massage.
  Other Names: reflection

SUMMARY:
The purpose of this study is to determine how parents of children with cancer rate a parent-delivered massage therapy educational program for usability and satisfaction, and if massage therapy, provided by parents to their child with cancer, reduce symptoms of anxiety and depression in the child, and parenting stress in the parent.

DETAILED DESCRIPTION:
In Canadian children aged 0-19, the number of new cancer cases from 1997-2001 was on average 1,285 children per year for a total of 6,427 children over a five year period. Individual and family responses to a child's or adolescent's cancer diagnosis and treatment include psychological, sociocultural and biological dimensions. Parents of children with cancer can experience severe emotional distress including anxiety and depression. Parents require support and skills to reduce their own anxiety and distress and to help alleviate suffering in their children.

This is a two-phase research project: phase I: development of a standardized educational intervention on video/DVD to teach parents how to massage their child with cancer; phase II: test the feasibility of the developed intervention with children with cancer and their parents. A total of 24 parents and their children with cancer who are under the care of the paediatric oncology units at the Stollery Children's Hospital (Edmonton) will be recruited for the study.

It is hypothesized that this research on an educational program in parent-delivered massage therapy will directly improve the lives of children with cancer and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 18 years
* Children with a life expectancy of at least 12 weeks
* Children who are currently receiving active cancer care

Exclusion Criteria:

* Children under the age of 6
* Children with a life expectancy of less than 12 weeks
* Children not currently receiving active cancer care

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
To test the feasibility of the educational intervention in parent-delivered massage for children undergoing treatment for cancer at a paediatric oncology centre, to guide sample size estimation for a future randomized trial. | Period of study

SECONDARY OUTCOMES:
My Story | Week 6
Memorial Symptom Assessment Scale | 0, 6, 12 weeks
Pediatric Inventory for Parents | 0, 6, 12 weeks
Stait-Trait Anxiety Inventory for Adults | 0, 6, 12 weeks
The Center for Epidemiologic Studies Depression (CES-D) Scale | 0, 6, 12 weeks
State-Trait Anxiety Inventory for Children | 0, 6, 12 weeks
Parent Journals | Weekly for 6 weeks
Child Journals | Weekly for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Trish Dryden, RMT, M.Ed, Principal Investigator — Applied Research Centre, Centennial College; Sabine Moritz, Dipl. Biol., M.Sc, Principal Investigator — Canadian Institute of Natural and Integrative Medicine; Sunita Vohra, MD, FRCPC, M.Sc, Principal Investigator — Stollery Children's Hospital & University of Alberta; Dawn Davies, MD, FRCPC, Principal Investigator — Stollery Children's Hospital; Adrienne D Witol, Psy.D., C.Psych, Principal Investigator — Stollery Children's Hospital; Andrea M Laizner, RN, Ph.D, Principal Investigator — Centre de recherché Hôpital Sainte-Justine CHU Mère-Enfant & McGill University Health Centre; Lyse Lussier, Principal Investigator — Le Phare enfants et familles; Janet Kahn, LMT, Ph.D., Principal Investigator — University of Vermont; Amanda Baskwill, RMT, Principal Investigator — Centennial College; Linda Curcher, CCRP, Principal Investigator — Stollery Children's Hospital; Elizabeth Barberree, RMT, Principal Investigator — Massage Therapist Association of Alberta (MTAA)
Locations (2):
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Centennial College, Toronto, Ontario

REFERENCES:
- [Background] Moore IM. Advancing biobehavioral research in childhood cancer. J Pediatr Oncol Nurs. 2004 May-Jun;21(3):128-31. doi: 10.1177/1043454204264400. PMID 15296039
- [Background] Boman K, Lindahl A, Bjork O. Disease-related distress in parents of children with cancer at various stages after the time of diagnosis. Acta Oncol. 2003;42(2):137-46. doi: 10.1080/02841860310004995. PMID 12801132
- [Background] Trask PC, Paterson AG, Trask CL, Bares CB, Birt J, Maan C. Parent and adolescent adjustment to pediatric cancer: associations with coping, social support, and family function. J Pediatr Oncol Nurs. 2003 Jan-Feb;20(1):36-47. doi: 10.1053/jpon.2003.5. PMID 12569433
- [Background] MacDonald G. Massage as a respite intervention for primary caregivers. Am J Hosp Palliat Care. 1998 Jan-Feb;15(1):43-7. doi: 10.1177/104990919801500109. PMID 9468978
- [Background] Cavusoglu H. Depression in children with cancer. J Pediatr Nurs. 2001 Oct;16(5):380-5. doi: 10.1053/jpdn.2001.0000. PMID 11598872
- [Background] Moyer CA, Rounds J, Hannum JW. A meta-analysis of massage therapy research. Psychol Bull. 2004 Jan;130(1):3-18. doi: 10.1037/0033-2909.130.1.3. PMID 14717648
- [Background] Cassileth BR, Vickers AJ. Massage therapy for symptom control: outcome study at a major cancer center. J Pain Symptom Manage. 2004 Sep;28(3):244-9. doi: 10.1016/j.jpainsymman.2003.12.016. PMID 15336336
- [Background] Field T, Cullen C, Diego M, Hernandez-Reif M, Sprinz P, Beebe K, Kissel B, Bango-Sanchez V. Leukemia immune changes following massage therapy. Journal of Bodywork & Movement Therapies 5(4): 271-274, 2001.
- [Background] Laizner AM, Lussier L. Massage provides comfort to children with cancer: the child's perspective. Journal of Complementary & Integrative Medicine 2(1): 34, 2005
- [Background] Fellowes D, Barnes K, Wilkinson S. Aromatherapy and massage for symptom relief in patients with cancer. Cochrane Database Syst Rev. 2004;(2):CD002287. doi: 10.1002/14651858.CD002287.pub2. PMID 15106172
- [Background] Laizner AM, Lussier L. Massage program relives suffering for parents while provides comfort for children. Journal of Complementary & Integrative Medicine 2(1): 35, 2005.
- [Background] Wilkinson S, Aldridge J, Salmon I, Cain E, Wilson B. An evaluation of aromatherapy massage in palliative care. Palliat Med. 1999 Sep;13(5):409-17. doi: 10.1191/026921699678148345. PMID 10659113
- [Background] Goodfellow LM. The effects of therapeutic back massage on psychophysiologic variables and immune function in spouses of patients with cancer. Nurs Res. 2003 Sep-Oct;52(5):318-28. doi: 10.1097/00006199-200309000-00006. PMID 14501546
- [Background] Rexilius SJ, Mundt C, Erickson Megel M, Agrawal S. Therapeutic effects of massage therapy and handling touch on caregivers of patients undergoing autologous hematopoietic stem cell transplant. Oncol Nurs Forum. 2002 Apr;29(3):E35-44. doi: 10.1188/02.ONF.E35-E44. PMID 11979292
- [Background] Bold J, Leis A. Unconventional therapy use among children with cancer in Saskatchewan. J Pediatr Oncol Nurs. 2001 Jan-Feb;18(1):16-25. doi: 10.1177/104345420101800103. PMID 11172406
- [Background] Kazak AE. Evidence-based interventions for survivors of childhood cancer and their families. J Pediatr Psychol. 2005 Jan-Feb;30(1):29-39. doi: 10.1093/jpepsy/jsi013. PMID 15610982
- [Background] Chambers B, Cheun A, Gifford R, Madden N. Achievement effects of embedded multimedia in a success for all reading program. Success for All Foundation (Grant No. REC 0115659): John Hopkins, 2004.
- [Background] Gecsedi RA. Massage therapy for patients with cancer. Clin J Oncol Nurs. 2002 Jan-Feb;6(1):52-4. doi: 10.1188/02.CJON.52-54. PMID 11842490
- [Background] Billhult A, Dahlberg K. A meaningful relief from suffering experiences of massage in cancer care. Cancer Nurs. 2001 Jun;24(3):180-4. PMID 11409061
- [Background] Forchuk C, Baruth P, Prendergast M, Holliday R, Bareham R, Brimner S, Schulz V, Chan YC, Yammine N. Postoperative arm massage: a support for women with lymph node dissection. Cancer Nurs. 2004 Jan-Feb;27(1):25-33. doi: 10.1097/00002820-200401000-00004. PMID 15108949
- [Background] Post-White J, Hawks RG. Complementary and alternative medicine in pediatric oncology. Semin Oncol Nurs. 2005 May;21(2):107-14; discussion 115-24. doi: 10.1016/j.soncn.2004.12.007. PMID 15991661
- [Background] Santo A, Laizner AM, Shohet L. Exploring the value of audiotapes for health literacy: a systematic review. Patient Educ Couns. 2005 Sep;58(3):235-43. doi: 10.1016/j.pec.2004.07.001. PMID 16054796
- [Background] Phipps S, Dunavant M, Gray E, Rai SN. Massage therapy in children undergoing hematopoietic stem cell transplant: results of a pilot trial. Journal of Cancer Integrated Medicine 3: 62-70, 2005.
- [Background] Cherkin DC, Sherman KJ, Deyo RA, Shekelle PG. A review of the evidence for the effectiveness, safety, and cost of acupuncture, massage therapy, and spinal manipulation for back pain. Ann Intern Med. 2003 Jun 3;138(11):898-906. doi: 10.7326/0003-4819-138-11-200306030-00011. PMID 12779300
- [Background] Furlan AD, Brosseau L, Imamura M, Irvin E. Massage for low-back pain: a systematic review within the framework of the Cochrane Collaboration Back Review Group. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1896-910. doi: 10.1097/00007632-200209010-00017. PMID 12221356
- [Background] Curties D. Massage therapy and cancer. Moncton, NB: Curties-Overzet Publications, 1988.
- [Background] Walton, T. Contraindications to massage part IV: clinical thinking and cancer. Massage Therapy Journal 39(3): 66-83, 2000.
- [Background] Field T, Hernandez-Reif M, Quintino O, Schanberg S, Kuhn C. Elder retired volunteers benefit from giving massage therapy to infants. Journal of Applied Gerontology 17(2): 229-239, 1998.
- [Background] Spielberger CD, Gorsuch RC, Lushene RE. The State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press, 1970.
- [Background] Spielberger CD, Edwards CD, Lushene RE, Montuori J, Platzek D. STAIC preliminary manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press Inc., 1973.
- [Background] Collins JJ, Byrnes ME, Dunkel IJ, Lapin J, Nadel T, Thaler HT, Polyak T, Rapkin B, Portenoy RK. The measurement of symptoms in children with cancer. J Pain Symptom Manage. 2000 May;19(5):363-77. doi: 10.1016/s0885-3924(00)00127-5. PMID 10869877
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Applied Psychogical Measure 1: 385-401, 1977.
- [Background] Streisand R, Braniecki S, Tercyak KP, Kazak AE. Childhood illness-related parenting stress: the pediatric inventory for parents. J Pediatr Psychol. 2001 Apr-May;26(3):155-62. doi: 10.1093/jpepsy/26.3.155. PMID 11259517
- [Background] Cresswell JW. Qualitative inquiry and research design: Choosing among five traditions. Thousand Oaks, Sage, 1998.
- See also: Leucan - Massage d'espoir — http://leucan.qc.ca/en
- See also: College of Massage Therapists of Ontario — http://www.cmto.com/index.html